CLINICAL TRIAL: NCT01867034
Title: Soluble Receptors for Advanced Glycation End-Products to Predict the Type of Stent Implant
Brief Title: Soluble Receptors for Advanced Glycation End-Products and PCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5516
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2012-03

CONDITIONS: Acute Coronary Syndrome
Keywords: non ST segment myocardial infarction
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bare Metal stent (Active Comparator): Stent that has not been impregnated with an anti-restenotic drug
  Interventions: Other: Bare Metal Stent
- Drug Eluting Stent (Active Comparator): Stent that has been impregnated with an anti-restenotic drug
  Interventions: Other: Drug Eluting Stent

INTERVENTIONS:
Other: Drug Eluting Stent — Comparison of two stents to see which results in best outcome.
  Arms: Drug Eluting Stent
Other: Bare Metal Stent
  Arms: Bare Metal stent

SUMMARY:
It is hypothesized that patients with low pre-PCI serum levels of sRAGE should receive DES implantation and/ or procedures taken to increase serum levels of sRAGE and/ or decrease the serum levels of AGE.

The purpose of this pilot study is to afford invasive cardiologists with additional evidenced based information to guide their decision as to which patients should receive a BMS or DES for coronary implantation.

The objectives of the study are to determine whether or not:

1. Patients with low pre-PCI serum levels of sRAGE who receive bare metal stents develop restenosis
2. Patients with high pre-PCI serum levels of sRAGE who receive bare metal stents will have reduced risk of the development of restenosis
3. Patients with low pre-PCI serum levels of sRAGE who receive drug eluting stents will have an increased risk of the development of restenosis

DETAILED DESCRIPTION:
Advanced glycation end products (AGE) are irreversible adducts formed from the non-enzymatic glycation and oxidation of proteins, lipids and nucleic acids. 1-4 AGE interacts with three types of cell receptors for advanced glycation end products (RAGE) namely full-length RAGE, N-truncated and C-truncated soluble receptors for AGE (sRAGE). The interaction of full-length RAGE with AGE increases the expression of adhesion molecules, including soluble vascular cell adhesion molecule-1 (sVCAM-1) and the cytokine tumor necrosis factor-α (TNF- α) activation of nuclear factor kappa B (NFκB) which in turn increases the expression of proinflammatory genes for adhesion molecules and cytokines, and the generation of reactive oxygen species (ROS). The function of N-truncated RAGE is poorly understood. sRAGE is not membrane bound and circulates in the plasma. Acting as a decoy for RAGE ligands (AGE), sRAGE competes with full-length RAGE for ligand binding. Consequently, sRAGE plays a protective role by preventing activation of full-length RAGE.

Adhesion molecules, cytokines, and ROS are involved in the development and progression of atherosclerosis and lesion instability. The AGE and RAGE axis is involved in the development atherosclerosis in diabetes. Balloon injury in carotid artery and endothelial denudation in animal models increases the levels of RAGE and AGE in the arterial wall and produce neointimal hyperplasia. Treatment with sRAGE in animal models reduces neointimal growth, decreases smooth muscle cell proliferation and migration, and expression of extracellular matrix. sRAGE reduces the atherosclerotic lesions in Apo-E -/- mice and this effect is associated with a decrease in aortic VCAM-1 and tissue factor.

Recently, we have demonstrated that the levels of serum sRAGE are lower while the serum levels of AGE, sVCAM-1 and TNF-α are higher in subjects with NSTEMI as compared to healthy controls 31. Furthermore, we have shown that the NSTEMI patients, who underwent PCI with BMS implantation and developed post-PCI restenosis after six-months, had lower serum levels of sRAGE as compared to those who did not 30. In the proposed study we expect to find that all patients with very low levels of serum sRAGE receiving either a BMS develop post-PCI restenosis while patients with very low serum levels of sRAGE receiving DES will increased rate of post-PCI restenosis. In addition, those patients with high levels of sRAGE who receive either BMS or DES will have a reduced rate of restenosis.

This study has clinical significance because in our previous study (McNair et al, 2010), we demonstrated that low serum levels of sRAGE are associated with 100% restenosis following BMS implantation. In these situations DES implantation will be highly beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NSTEMI
* Discrete denovo localized lesions in single or multiple vessel
* Non-diabetic
* EF> 40%
* Patients willing to come back for a follow-up angiogram 6 months post -PCI

Exclusion Criteria:

* The reference diameter artery less than 2.5 mm in diameter
* STEMI
* Post-coronary artery bypass graft surgery
* Diabetic
* Coexisting inflammatory diseases
* Coexisting valvular disease
* Patients with a history of substance abuse

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
sRAGE | 6-months
  The serum levels of sRAGE will be determined at six months.

SECONDARY OUTCOMES:
coronary restenosis | 6-months
  The patient will have a followup angiogram to determine if restenosis is present.

CONTACTS AND LOCATIONS:
Overall Officials: Erick McNair, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada